CLINICAL TRIAL: NCT00944996
Title: Assessment of PACAP-BDNF Signaling System Involvement in Etiology and Treatment of Major Depression
Brief Title: Assessment of Pituitary Adenylate Cyclase Activating Polypeptide-Brain Derived Neurotrophic Factor (PACAP-BDNF) Signaling System Involvement in Etiology and Treatment of Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tirat Carmel Mental Health Center (Other Government)
Collaborators: University of Michigan (Other); Ariel University (Other); The Nazareth Hospital, Israel (Other)
Responsible Party: Principal Investigator, Anatoly Dr. Kreinin, Director of Psychiatric Department, Tirat Carmel Mental Health Center
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: akparl08; 920080174; 040-2008
Record Dates: First submitted 2009-07-19; First posted 2009-07-23 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Major Depression
Keywords: PACAP (Pituitary Adenylate Cyclase Activating Polypeptide); Major Depression; Receptors; Gene polymorphism; PACAP signaling system; Etiology of major depression; Mechanism of antidepressants action; PACAP receptors gene polymorphism; Pathogenesis of major depression; Responsiveness to the antidepressant drugs
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Selective Serotonin Reuptake Inhibitors; Serotonin and Noradrenaline Reuptake Inhibitors; Paroxetine; Fluoxetine; Sertraline; Escitalopram; Citalopram; Venlafaxine Hydrochloride; Clomipramine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- antidepressant (Active Comparator)
  Interventions: Drug: SSRI; SNRI; TCA
- Healthy volunteers (No Intervention)

INTERVENTIONS:
Drug: SSRI; SNRI; TCA — Tablets or Pills, 1 or 2 per day, more than 2 month
  Other Names: paroxetine, fluoxetine, sertraline, escitalopram, citalopram; mirtrazapine, venlafaxine; anafranil
  Arms: antidepressant

SUMMARY:
The neuropeptide Pituitary Adenylate Cyclase Activating Polypeptide (PACAP) and its receptors PAC1 and VPAC2 are widely expressed in the nervous system. The investigators found that PACAP treatment of neuronal cell cultures increases expression of Brain Derived Neurotrophic Factor (BDNF) that plays an important role in the etiology of psychiatric disorders and action of antidepressants. For the first time, the investigators demonstrated that treatment by Paroxetine and Citalopram significantly decreases PAC1 and VPAC2 and upregulates PACAP mRNA expression, whereas Imipramine shows an opposite effect. Moreover, PACAP, PAC1 and VPAC2 expression is highly correlated with BDNF expression. Their in vivo studies show that Imipramine reduces BDNF and increases PAC1 mRNA expression in murine hippocampus, suggesting that antidepressants may affect neuronal plasticity through PACAP-BDNF interactions. Based on their observations in experimental systems, the investigators hypothesize that PACAP signaling system may be involved in the etiology of depression and mechanism of antidepressant action. The investigators will evaluate this hypothesis by examining serum PACAP levels, effect of antidepressants on PACAP levels, and gene polymorphisms of PACAP and its receptors in major depressive disorder patients. This study will enhance the investigators' understanding of PACAP's role in the etiology of depression and antidepressant treatment and will provide a basis to evaluate PACAP pathway as a potential target for diagnostics and novel antidepressants drug discovery.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18-65 age old
2. Patients with DSM-IV (or/and ICD-10) diagnosis MDD
3. Volunteers without DSM-IV (or/and ICD-10) diagnosis MDD
4. For patients with DSM-IV (or/and ICD-10) diagnosis MDD minimum 2 weeks free from benzodiazepines, mood stabilizers and neuroleptics.
5. All patients from MDD group treatment only by SSRI antidepressant medications.

Exclusion Criteria:

1. MDD with Co-morbidity
2. Alcohol and drug use less than 1 month before the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Measurements of PACAP and BDNF serum levels | Blood samples will be collected at the study base line, two and three weeks after that and at the study end point (8 weeks after study initiation)
Analysis of genetic variants of PACAP and PAC1 coding and regulatory regions | Blood samples will be collected at the study base line, two and three weeks after that and at the study end point (8 weeks after study initiation)

CONTACTS AND LOCATIONS:
Overall Officials: Anatoly Kreinin, MD, PhD, Study Chair — The Bruce and Ruth Rappaport Faculty of Medicine, Technion, Haifa; Albert Pinhasov, PhD, Principal Investigator — Department of Molecular Biology at Ariel University Center; Leon Raskin, PhD, Principal Investigator — University of Michigan; Kamal Farhat, MD, Principal Investigator — The Nazareth Hospital-EMMS; Joseph Farah, MD, Principal Investigator — The Nazareth Hospital-EMMS; Klaudia Rybalksy, MD, Principal Investigator — The Nazareth Hospital-EMMS
Locations (1):
- Tirat Carmel Mental Health Center, Tirat Hacarmel, Israel